CLINICAL TRIAL: NCT03923686
Title: Endoscopic Ultrasound-guided Drainage Using Lumen-apposing Metal Stent With or Without Coaxial Plastic Stent for Treatment of Walled-off Pancreatic Necrosis: a Prospective Randomised Study
Brief Title: Lumen-apposing Metal Stent With or Without Coaxial Plastic Stent for Treatment of Walled-off Pancreatic Necrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Petr Vanek, Principal Investigator, Palacky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNOL 2IK 001
Record Dates: First submitted 2019-04-12; First posted 2019-04-22 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Pancreatitis, Acute Necrotizing; Walled Off Necrosis
Keywords: Walled off necrosis; Acute pancreatitis; Necrotizing pancreatitis; Endoscopic drainage; Lumen apposing metal stents; Double pigtail plastic stent
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis

STUDY DESIGN:
Intervention Model Description: a prospective randomized cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAMS plus DPS (Experimental): Endoscopic ultrasound-guided (EUS) transmural drainage of walled-off pancreatic necrosis (WON) using lumen-apposing metal stent (LAMS) with coaxial double-pigtail plastic stent (DPS).
  Interventions: Procedure: EUS-guided drainage using LAMS with DPS
- LAMS alone (Active Comparator): Endoscopic ultrasound-guided (EUS) transmural drainage of walled-off pancreatic necrosis (WON) using lumen-apposing metal stent (LAMS) alone.
  Interventions: Procedure: EUS-guided drainage using LAMS alone

INTERVENTIONS:
Procedure: EUS-guided drainage using LAMS with DPS — Endoscopic ultrasound-guided drainage using lumen-apposing metal stent with coaxial plastic stent in the treatment of walled-off pancreatic necrosis.
  Arms: LAMS plus DPS
Procedure: EUS-guided drainage using LAMS alone — Endoscopic ultrasound-guided drainage using lumen-apposing metal stent without coaxial plastic stent in the treatment of walled-off pancreatic necrosis.
  Arms: LAMS alone

SUMMARY:
A prospective randomized cohort study to compare whether the placement of a double-pigtail plastic stent (DPS) within a lumen-apposing metal stent (LAMS) may improve the efficacy and safety of endoscopic ultrasound guided transmural drainage of walled-off pancreatic necrosis (WON) and thus prevent potential adverse events related to LAMS insertion.

DETAILED DESCRIPTION:
The aim of the study is to compare endoscopic ultrasound guided transmural drainage using lumen-apposing metal stent with (1.) or without (2.) coaxial plastic stent in the management of walled-off pancreatic necrosis. The usage of LAMS has been evaluated as a safe and effective method for the drainage of walled-off pancreatic necrosis in various studies. However, complications such as bleeding, infection due to stent obstruction, stent migration, or buried stent syndrome have been reported. A preventive measure to minimize adverse events related to LAMS insertion by means of placing an anchoring DPS through the LAMS have been suggested but there has been no prospective randomized study to assess the utility of such measure to date.

The study is to be conducted at a tertiary institution with an expertise in treating hepato-pancreato-biliary diseases. The main timeframe of the study is 3 weeks following LAMS insertion with or without DPS. All LAMS will be extracted 3 weeks after the initial procedure. The extraction will be preceded by a CT scan of the abdomen to assess whether the DPS needs to be left in place/ inserted in patients with incomplete resolution of the collection. In addition, material from the collection will be collected for cultivation at every endoscopic intervention to assess colonization by microbial flora over time. All patients will be closely followed with clinical, laboratory, and radiological assessment for 12 months in total.

Our experience has shown failure of the (2.) method in 70 % of patients so far. Assuming a clinically significant difference to be a reduction to 40 % in failed patients using the (1) method, the required study population size was calculated to 62 patients (31 in both arms) by power analysis (at standard alpha and beta values). The final number was set to 70 as a safety measure.

ELIGIBILITY:
Inclusion Criteria:

* walled-off pancreatic necrosis (WON) indicated for endoscopical drainage
* signed informed consent form

Exclusion Criteria:

* patient disagreement with the study
* types of collections other than WON
* drainage with stents other than LAMS
* previous attempts at drainage of WON
* severe coagulopathy or thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Failure of method | up to 1 month
  Defined as a necessity of re-intervention (endoscopic, surgical, percutaneous) within the period following LAMS insertion and before its planned extraction due to complications related to LAMS insertion and/or clinical deterioration.
Mortality | up to 12 months
  Overall mortality during subsequent follow-up

SECONDARY OUTCOMES:
Clinical success rate | up to 1 month
  Resolution of the collection and symptoms following endoscopic drainage with LAMS before its extraction.
Adverse events | up to 1 month
  Primarily complications caused by LAMS itself (bleeding due to vessel erosion, secondary infection due to stent obstruction, stent migration, buried stent syndrome).
Number of procedures | up to 1 month
  Number of forced endoscopic interventions (direct endoscopic necrosectomy, debridement, desobliteration, etc.) required to achieve resolution.
Hospital stay | up to 1 month
  Total length of hospital stay within the period following LAMS insertion until its extraction.
Recurrence rate | up to 12 months
  Recurrence of the collection accompanied by symptoms provided there had been previous clinical success with documented resolution of the collection by radiological studies.
Microbiological cultivation | up to 1 month
  Material from the collection will be collected at every endoscopic intervention (at least during insertion and extraction of LAMS) to assess colonization by microbial flora over time.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Vanek, MD, Principal Investigator — Assistant Professor, physician
Locations (1):
- University Hospital Olomouc, Second Department of Internal Medicine - Gastroenterology and Geriatrics, Olomouc, Czechia

REFERENCES:
- [Derived] Vanek P, Falt P, Vitek P, Zoundjiekpon V, Horinkova M, Zapletalova J, Lovecek M, Urban O. EUS-guided transluminal drainage using lumen-apposing metal stents with or without coaxial plastic stents for treatment of walled-off necrotizing pancreatitis: a prospective bicentric randomized controlled trial. Gastrointest Endosc. 2023 Jun;97(6):1070-1080. doi: 10.1016/j.gie.2022.12.026. Epub 2023 Jan 13. PMID 36646148